CLINICAL TRIAL: NCT06357936
Title: Nanofat Grafting as a Method of Treating Critical Limb Ischemia - Pilot, Prospective Randomised Blinded Trial
Brief Title: Nanofat Grafting as a Method of Treating Critical Limb Ischemia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Center of New Medical Technologies (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CNMT002
Record Dates: First submitted 2024-04-05; First posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Limb Ischemia
Keywords: Nano fat grafting; Critical limb ischemia; Autologous stem cells; Limb preservation
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nano fat grafting group (Experimental)
  Interventions: Procedure: nano-fat grafting in chronic limb ischaemia
- standard therapy group (Sham Comparator)
  Interventions: Procedure: sham comparator

INTERVENTIONS:
Procedure: nano-fat grafting in chronic limb ischaemia — The nano fat grafting procedure in the clinical trial involves the collection of adipose tissue under tumescent anesthesia, which is a technique to swell and firm the targeted area, through a separate puncture in the anterior abdominal wall. Following the collection, the adipose tissue undergoes a process of cannulation to prepare the nano fat. This prepared material is then injected into the tissues of the foot and leg using standard intramuscular injection needles. The injections are performed in various directions to ensure proper distribution of the nano fat. This method does not require additional drug therapy. It leverages the natural growth factors and stem cells present in adipose tissue, aiming to improve blood flow and tissue regeneration in limbs affected by critical ischemia. The unique aspect of this treatment is its focus on using autologous materials, minimizing the risk of rejection and side effects associated with foreign substances.
  Arms: nano fat grafting group
Procedure: sham comparator — For the clinical trial, a sham procedure would be designed to mimic the nano fat grafting without providing the actual therapeutic intervention. This involve the patient undergoing a similar process with tumescent anesthesia and making a puncture on the anterior abdominal wall. However, instead of harvesting adipose tissue and preparing nano fat, a placebo solution (such as saline) would be injected using the same intramuscular injection technique. The aim of this sham comparator is to assess the psychological and physiological effects of the nano fat grafting procedure itself, by eliminating the potential therapeutic benefits of the nano fat.
  Arms: standard therapy group

SUMMARY:
This clinical trial will investigate nano fat grafting as a method for treating critical limb ischemia. The method involves the collection of adipose tissue under tumescent anesthesia through a separate incision in the anterior abdominal wall, followed by preparation and injection of nano fat into the tissues of the foot and leg without additional drug therapy. The novelty of this method lies in the use of autologous stem cells and growth factors, differing from current treatments like neovasculgen, which is a plasmid DNA-based treatment. The trial aims to assess the safety and effectiveness of nano fat grafting, including pain relief, the frequency of intraoperative complications, increased distance of pain-free walking, limb preservation, and mortality rates.

The trial will involve patients with diagnosed occlusive lesions of the femoral-popliteal-tibial segment and chronic ischemia of III-IV degree according to Fontaine and 5-6 categories according to Rutherford, excluding those with contraindications for surgical intervention on the femoral-popliteal-tibial segment, chronic heart failure of III-IV NYHA class, severe liver or kidney failure, among others.

The study design includes preoperative examinations, hospital phase activities including the surgery and post-operative assessments, and follow-up visits at 6 and 12 months post-operation to evaluate the method's safety, complications, and effectiveness based on various parameters like pain, trophic disturbances, and limb ischemia severity.

Statistical methods will involve quantitative data presented as mean ± standard deviation, with qualitative traits compared using the Chi-square test or Fisher's exact test. The planned patient number is 40, aiming to demonstrate the effectiveness and safety of nano fat grafting for critical limb ischemia treatment compared to current treatments.

ELIGIBILITY:
Inclusion Criteria:

* Patients with occlusive lesions of the femoral-popliteal-tibial segment.
* Chronic ischemia of the lower limbs of III-IV degree according to Fontaine and categories 5-6 according to Rutherford.
* Signed informed consent for participation in the clinical trial.

Exclusion Criteria:

* Absence of indications for surgical intervention on the femoral-popliteal-tibial segment.
* Patients refusing to participate in the clinical trial.
* Chronic heart failure of III-IV NYHA functional class.
* Chronic decompensated "pulmonary" heart.
* Severe liver or kidney failure (bilirubin >35 mmol/L, glomerular filtration rate <60 ml/min).
* Polivalent drug allergy.
* Malignant oncological diseases in the terminal stage with a life expectancy of less than 6 months.
* Acute cerebrovascular accident.
* Decompensated diseases of the endocrine organs (for diabetes, glycemia level more than 10 mmol/L).
* Pregnancy and lactation period.
* Inability to undergo examinations at control points.
* Refusal to sign informed consent for participation in the clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-04-20 (Estimated); Primary Completion 2024-11-20 (Estimated); Study Completion 2025-02-20 (Estimated)

PRIMARY OUTCOMES:
Percent of pain absence in experimental group | 12 months

SECONDARY OUTCOMES:
Number of any intraoperative complications | 12 months
Number of any inhospital complications | 12 months
Number of saved limbs | 12 months
Percent change in visual analog pain score (VAS) change | 12 months
  The Visual Analogue Scale (VAS) is a straightforward, tool for measuring pain intensity or other subjective experiences that are difficult to quantify, such as fatigue or nausea. It consists of a straight line, usually 10 centimeters (100 millimeters) long, anchored by two descriptors defining the extremes of the experience being measured (e.g., "no pain" on one end and "worst imaginable pain" on the other for pain measurement).. The result is typically recorded in millimeters, with scores ranging from 0 to 100, where 0 represents one extreme (e.g., no pain) and 100 represents the other (e.g., worst imaginable pain).

CONTACTS AND LOCATIONS:
Locations (1):
- Center of New Medical Technologies, Novosibirsk, Novosibirsk Oblast, Russia